CLINICAL TRIAL: NCT01007981
Title: A Novel Echocardiography Modality to Assess Left Ventricular Dyssynchrony: Hemodynamic Assessment by 4D Segmental Ejection Fraction
Brief Title: A Novel Echocardiography Modality to Assess Left Ventricular Dyssynchrony
Status: Withdrawn | Type: Observational
Why Stopped: investigator left the institution
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: 1124400
Record Dates: First submitted 2009-11-04; First posted 2009-11-05 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CRT device: Patients with Cardiac Resynchronization Therapy(CRT) device implanted in the last 5 years will be studied by the new echo modality.Study doesn't involve acute device implantation.

SUMMARY:
The investigators hypothesize that the relation between mechanical and hemodynamic left ventricular dyssynchrony might better predict response to Cardiac Resynchronization Device(CRT) than currently existing echo indices.

DETAILED DESCRIPTION:
Cardiac resynchronization therapy is emerging to be a highly effective treatment option for selected patients with symptomatic congestive heart failure on optimal medical therapy and evidence of left ventricular (LV) conduction delay and contraction dyssynchrony. It can improve quality of life and results in better survival in this selected group of patients. However, patients have different responses to CRT, and up to 30% of those implanted show no response at all. Ongoing trials, whether prospective or retrospective, have been trying to define best predictors of response to CRT and to measure ventricular dyssynchrony. Despite this, no single echo criterion to date can predict successful CRT over current guidelines.

In this study, we propose to compare LV muscle mechanical dyssynchrony assessment by speckle tracking to hemodynamic dyssynchrony assessment by 4D segmental ejection fraction (EF), a novel modality brought recently by University of Missouri Echocardiography laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac Resynchronization Therapy(CRT) device implanted in the last 5 years.

Exclusion Criteria:

* Acute decompensated congestive heart failure.
* chronic permanent atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed in cardiology clinic will be included.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
4D echo is the best modality to measure systolic dyssynchrony index | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Firas H El Sabbagh, MD, Principal Investigator — University of Missouri-Columbia

IPD SHARING:
Plan to Share IPD: No